CLINICAL TRIAL: NCT02168985
Title: Impact Evaluation for the Faithful House Program in Reducing Violence in Families in Which Couples Are Discordant or HIV/AIDS Positive in Arusha Region, in Tanzania
Brief Title: Impact Evaluation Study of The Faithful House Programme on Violence Reduction in Families
Acronym: TFHEVAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Savannas Forever Tanzania (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); Arusha Lutheran Medical Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFTZ-C&VECF
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Child Maltreatment
Keywords: Child violence; HIV AIDS conflicted couples; Intimate partner violence; Tanzania; Marriage counseling; Child maltreatment; Couples communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attend TFH Program (Experimental): Couples attend the three-day Faithful House Training program immediately
  Interventions: Behavioral: TFH program
- Wait-listed for TFH Program (No Intervention): Couples attend The Faithful House program three-months after the initial group

INTERVENTIONS:
Behavioral: TFH program — The Faithful House (TFH), is a three-day faith-based skills-building curriculum. The curriculum aims to increase household resilience by strengthening families and couples' relationships through enhanced couple communication
  Other Names: The Faithful House Training (TFH) Program
  Arms: Attend TFH Program

SUMMARY:
The Faithful House (TFH), is a 3-day faith-based skills-building curriculum which aims to increase household resilience by strengthening families. TFH draws on improved communication and conflict resolution skill building and the individual's faith-values as a catalyst for transformation in attitudes regarding gender roles in care giving and the use of violence in the home. The study hypothesis is that couples who complete the Faithful House Programme will demonstrate increased communication skills with their spouses and children, which reduces the negative impact of family stress triggers and ultimately leads to a reduction of intimate partner violence witnessed by children as well as physical and emotional violence against children by parents.

The mixed methods study will include a Randomized Control Trial (RCT) of HIV/AIDS infected or conflicted couples and a child in each household, focus group discussions (FGD) of men, women and children and key informant interviews of local experts in family violence and social protection service network providers.

DETAILED DESCRIPTION:
A mixed-method evaluation of The Faithful House is proposed. In the main, we will conduct a randomized control trial of the education program to determine treatment effect. We will also conduct semi-structured interviews and focus groups with stakeholders. This more qualitative work will be done in order to refine our program and evaluation and to assess the fidelity of the intervention and assess and unintended consequences. Informed consent will be sought from all prospective participants.

The source population is families that receive HIV care from Arusha Lutheran Medical Centre and Selian Hospital. Participation and related compliance is enhanced because subjects come to the hospital for HIV treatment. Couples with children ages 10 to 17 years will be recruited to participate in a Faithful House workshop and study by hospital volunteers. All patients attending the clinic during the recruiting period will be screened based on eligibility criteria. The list of patients screened will be checked against the clinic register to verify that all potential participants were screened and all eligible respondents were invited to participate in the workshop and study.

The list of recruited couples will be randomized to receive the intervention or to serve as the control arm. The control arm will be offered the intervention at the conclusion of the study. The goal is to have N=150 couples in the treatment arm and N=150 couples in the control arm. The rationale for the sample size is twofold. First, given the estimated variances from surveillance studies the sample size permits the estimates of small to moderate effect sizes at 80% power and 5% Type I error. In simple terms, the proposed evaluation is strongly powered to detect politically and clinically meaningful effects. Second, given time, budget, and patient flow characteristics, 300 couples is near the maximum of our capacity. Baseline measures will be taken via survey on all participants in a clinical setting about one month prior to beginning the education program. Post program measures will be taken in a clinical setting three months after the intervention is complete. A context-based pretest and post-test will be administered to only those in the treatment group on the first and last day of the intervention.

Gender and age specific surveys will be used to interview men, women and children and questions on self-reported violence will be included in women and children's questionnaires. Answers to questions on violence will be collected using non-verbal response cards to protect confidentiality and to assure respondents that enumerators will not know their responses.

Analyses will focus mainly on difference in estimates for the primary outcome measures of the self reported incidence by mothers and children (10-17) of acts of violence against women and children including child-witnessed violence in the past three months before the intervention and three months post intervention. Sub-group analysis by gender will be conducted. We will look at within group difference and between group differences. Retention will be assessed by comparing results from the pretest and post-test given on the first and last day of the intervention.

Secondary analyses on secondary outcomes such as parental attitudes toward violence and abuse and changes in intimate partner violence. We will examine the hypothesized theoretical links (e.g., mediation) between observed outcomes and program characteristics. A two-sample t-test will be used to look for differences in incidence of violence between the intervention and control groups. Multiple regression will be used to identify and examine predictor variables.

All data will be collected using electronic pads that contain self-checking logic within the questionnaire. Should missing data exceed 10%; multiple imputation procedures will be employed. However, our experience in similar studies is that imputation was not required because our fielding processes led to very high completions in the field.

Study instruments will include before focus group discussions (FGD) prior to the intervention, baseline, before and after workshop tests, three-month follow-up interviews, and post analysis FGD. Where possible, questions from other family and child violence studies will be utilized to allow for inter-study comparisons, especially focusing on evaluation studies of other The Faith House education programs and on the Violence Against Children in Tanzania National Survey conducted in 2009. All differences will be reported at a p <0.05. Data analysis will be completed using Stata v12. Importantly, we will also conduct a qualitative comparison of our outcome measures with published surveillance estimates in order to learn more about our source population and the potential impact of our program on the area if scaled up. As mentioned above, we will conduct interview and focus groups to improve program development, assess the fidelity of the implementation, and potential unintended consequences. Indeed, on-going study results will be monitored and a priori stopping rules assessed.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female partners in an HIV AIDS conflicted couple
* Has at least one child age 10 to 17 years living in couple's household

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-10 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of violence against or witnessed by children insults, and threats of physical harm and abandonment in the past three months and similar violent acts between partners that are observed by their children ages 10-17. | Baseline and three months after couples attend seminar
  Change in self-reported incidence by parents and children (10-17) of acts of physical and emotional violence against children such as kicking, hitting, verbal insults, and threats of physical harm and abandonment and similar violent acts between partners that are observed by their children ages 10-17 years at baseline and three-months after couples attend seminar.

SECONDARY OUTCOMES:
Attitudes about violence | Baseline and three months after seminar
  The study will measure changes in men, women's and children (age 10-17) attitudes related to the use of emotional and physical violence using self-reported ratings of agreement using agreement (yes/no) or (strongly disagree, disagree, neither agree nor disagree, agree and strongly agree) on statements about the acceptability of violence in different situations such as infidelity, burning food, disobedience. Respondents survey at baseline and three months after seminar.

CONTACTS AND LOCATIONS:
Overall Officials: Susan M James, MBA, Principal Investigator — Savannas Forever Tanzania; Sarah Milder, MPH, Principal Investigator — Arundel Street Consulting; Bernard J Ngowi, MD PhD, Principal Investigator — National Institute for Medical Research
Locations (1):
- Arusha Lutheran Medical Centre, Arusha, Arusha, Tanzania

REFERENCES:
- See also: Savannas Forever Tanzania is a research organization in Tanzania — http://sftz.org
- See also: National Institute for Medical Research — http://www.nimr.or.tz
- See also: Selian Hospital and Selian Aids Control Programme — http://selianlh.habari.co.tz/